CLINICAL TRIAL: NCT07019207
Title: The Effect of Virtual Reality-Based Dual-Task Training on Cognition, Cortical Activation, and Functional Level in Patients With Spinal Cord Injury
Brief Title: Virtual Reality Dual Task Training in SCI: Effects on Cognition and Cortical Activation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeUni-OCAKMAK-001
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: Dual-task; Virtual Reality; Cognition; Spinal Cord Injuries; Cortical Activation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria will be randomly assigned to one of three groups: a VR-based dual-task training with motor imagery group, a VR-based dual-task training without motor imagery group and a control group. Each arm will receive a distinct intervention protocol concurrently over the same study period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-Based Dual-Task Training with Motor Imagery Group (Experimental): In addition to the treatment to be applied to the participants in this group for upper extremity strengthening, they will complete a dual-task game designed by the researchers and involving cognitive-motor activity-based motor imagery that can be used with virtual reality glasses. Patients in this group will perform motor tasks during the game by seeing themselves standing and walking. Simultaneously with the game, an environment where the wheelchair can move safely will be created to prevent symptoms such as dizziness and nausea in patients and the wheelchair will be moved by the researcher in this environment. Participants will perform the game consisting of 3 different stages during one session. The motor task will be the same in all phases, the cognitive task will change.
  Interventions: Behavioral: VR-Based Dual-Task Training with Motor Imagery
- VR-Based Dual-Task Training without Motor Imagery Group (Experimental): Participants in this group will perform upper extremity strengthening exercises, similar to the other groups. Additionally, they will engage in a game that is identical in design to that used in the first group, but without incorporating motor imagery. The key distinction from the first group is that during the game, participants will achieve mobility via a wheelchair instead of performing the motor task of walking. Consequently, no motor imagery related to walking will be involved. To prevent symptoms such as dizziness and nausea during the game, a safe environment will be created in which the wheelchair can move securely. The wheelchair will be moved within this environment by the researcher. The main difference between the stages will be the progressively increasing difficulty of the cognitive tasks.
  Interventions: Behavioral: VR-Based Dual-Task Training without Motor Imagery
- Control Group (Active Comparator): This group is designated as the control group. Participants will receive only standard rehabilitation interventions, consisting of resistance band strengthening exercises based on proprioceptive neuromuscular facilitation (PNF) patterns and techniques commonly used in clinical practice.
  Interventions: Behavioral: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Behavioral: VR-Based Dual-Task Training with Motor Imagery — Participants will perform the game consisting of 3 different stages during one session. The motor task will include crossing the street between cars and walking on the sidewalk without hitting people. The difference between the stages will be the cognitive task, which becomes more difficult with each stage. The cognitive task in the first stage of the game will involve the colors that the patient will see and the simultaneous sound of the colors. The cognitive task in the second stage of the game will involve writing the names of some colors with black paint and reading them simultaneously. In the third stage of the game, the patient will see color names written with some colors. Every 5 seconds a new match will appear and the number of errors made during the matches will be recorded. In addition, upper extremity strengthening with PNF methods such as hold relaxation, rhythmic stabilization and repetitive stretches will be studied.
  Arms: VR-Based Dual-Task Training with Motor Imagery Group
Behavioral: VR-Based Dual-Task Training without Motor Imagery — The difference of this group from the first group is that they will see that they provide mobility with a wheelchair instead of walking, which is a motor task. In this case, there will be no motor imagery of walking. Simultaneously with the game, an environment where the wheelchair can move safely will be created in order to prevent symptoms such as dizziness and nausea in the patients and the wheelchair will be moved in this environment by the researcher. The difference between the stages will be the cognitive task that becomes more difficult at each stage and it will take a total of 20 minutes to complete all stages of the game. In addition, upper extremity strengthening will be practiced with PNF methods of hold and relax, rhythmic stabilization and repetitive stretches.
  Arms: VR-Based Dual-Task Training without Motor Imagery Group
Behavioral: Proprioceptive Neuromuscular Facilitation — The patients in the group will be applied only the resistance band strengthening methods including the upper extremity proprioceptive neuromuscular facilitation (PNF) patterns and methods applied as standard in rehabilitation. Strengthening will be worked on in all upper extremity PNF patterns using the resistance band with the PNF methods of hold-relax, rhythmic stabilization and repetitive stretching.
  Arms: Control Group

SUMMARY:
Spinal cord injury (SCI) is a severe neurological condition characterized by the loss of motor and sensory functions due to damage in the spinal cord or the nerves branching from it. Although studies investigating cognitive function after SCI are limited, it has been reported that up to 60% of individuals experience cognitive impairments. Because of impaired motor control, patients may need to invest more cognitive effort to perform even simple movements. This situation can negatively affect their ability to carry out multiple tasks at the same time and to respond effectively to environmental threats while walking, which may increase their risk of falling. Although the presence of cognitive changes after SCI is recognized in the literature, there are only a few studies examining the effects of rehabilitation on cortical activation, highlighting the need for innovative approaches to improve both motor and cognitive functions. The aim of this randomized controlled study is to investigate the effects of virtual reality (VR)-based dual-task training, both with and without motor imagery, on cortical activation, cognition, and functional level in individuals with SCI. Participants who meet the inclusion criteria will be recruited from the Turkish Spinal Cord Paralytics Association and will be randomly assigned to one of three groups: (1) a VR-based dual-task training group including motor imagery (n=15), (2) a VR-based dual-task training group without motor imagery (n=15), and (3) a control group (n=15). After obtaining informed consent and recording demographic data, pre-treatment (T0) and post-treatment (T1) assessments will be conducted. Cortical activation will be measured using functional near-infrared spectroscopy (fNIRS), grip strength with a Jamar hand dynamometer, upper extremity functional level with the Fugl-Meyer Assessment, sitting balance with the Modified Functional Reach Test, cognitive status with the Montreal Cognitive Assessment (MoCA), and occupational performance with the Canadian Occupational Performance Measure (COPM). Patient satisfaction and general health status will also be recorded. In addition to upper extremity strengthening exercises, patients in the VR groups will perform a cognitive-motor dual-task game developed by the researchers, which is played with VR glasses. The motor imagery group will complete the tasks while visualizing themselves standing and walking, while the other group will play the same game without walking imagery, from a wheelchair perspective. The game will involve motor tasks such as crossing the street between moving cars and walking on the sidewalk without bumping into people, as well as cognitive tasks based on the Stroop test, which will become progressively more difficult through three stages. Completing all stages will take approximately 20 minutes. Patients in the control group will only receive upper extremity strengthening exercises. The intervention will last for 12 sessions, conducted twice a week. The findings of this study are expected to emphasize the importance of simultaneous motor and cognitive rehabilitation in individuals with SCI and to contribute scientifically to the use of VR-supported innovative approaches in rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-60 years old
* Having full or partial paraplegia
* Having an injury level of T1 or below
* Having at least 90° active shoulder flexion and abduction
* Having at least 3 months since the injury

Exclusion Criteria:

* Musculoskeletal pain greater than 5 out of 10 on the Visual Analog Scale
* Patients who cannot sit in a chair for at least 30 minutes
* Presence of deformities or color changes in joints that prevent upper extremity movements
* Patients who have had fractures or operations on the upper extremity within the last 6 months
* History of head trauma
* Presence of a disease known to affect cognitive impairment
* Severe deafness, blindness or significant physical illnesses that cause communication disorders and prevent patients from participating in the study
* Presence of any known cardiovascular disease
* Conditions in which virtual reality glasses are contraindicated (epilepsy; vertigo and similar severe movement disorders)
* Patients with a history of stroke or progressive neurodegenerative disease
* Patients with neuromuscular disease
* Patients with uncontrolled epilepsy
* Concurrent participation in other studies or treatments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Cortical Hemodynamics (Functional Near-Infrared Spectroscopy) | Pre-treatment (Week 0) and after treatment (Week 6)
  A portable functional near-infrared spectroscopy (fNIRS) system (Brite MKIII, Artinis, The Netherlands) will be used to monitor hemodynamic changes during patients' cognitive tasks. Optode placement will be based on previous studies and Brodmann areas. Data will be simultaneously collected and analyzed using OxySoft software. The device includes ten emitters and eight detectors arranged in a 2 × 12 channel layout, covering cortical regions related to upper extremity representation. Channels will be symmetrically distributed across hemispheres. The emitter-detector distance will be set at 30 mm, and light wavelengths of 763 nm and 842 nm will be used. HbO₂ concentrations in regions of interest (PFC, SFC, SMA, and PMC) will be measured. ΔHbO₂, ΔHbR, and ΔHbT values will be recorded per channel as time-series data in units of μmol/L.
Upper Extremity Functional Level (Fugl-Meyer Motor Assessment Scale - Upper Extremity (FMA)) | Pre-treatment (Week 0) and after treatment (Week 6)
  The scale consists of five sections: motor function (upper and lower extremities), sensory function, balance, joint range of motion, and joint pain; however, the motor function assessment is the most commonly used section. It includes 33 items, each scored on a three-point ordinal scale based on the participant's ability to perform the task. For the upper extremity motor function, a participant can achieve a maximum score of 66. Higher scores indicate better motor function.
Cognition (Montreal Cognitive Assessment Test (MoCA)) | Pre-treatment (Week 0) and after treatment (Week 6)
  MoCA consists of nine subtests. It assesses multiple cognitive domains, including executive functions (e.g., trail making), visuospatial abilities (clock drawing task and three-dimensional cube copying), attention, concentration, working memory, language (e.g., a three-item naming task with low-familiarity animals), short-term memory, and orientation to time and place. These correspond to the following MoCA subtests: trail making, visuoconstructional skills, naming, attention, sentence repetition, verbal fluency, abstraction, delayed recall, and orientation. A score of 21 or higher on the scale is considered normal.
Sitting Balance (Modified Functional Reach Test) | Pre-treatment (Week 0) and after treatment (Week 6)
  The test is conducted with the individual seated in a standard wheelchair with footrests. The measuring rod is mounted on the wall at the level of the acromion process of the shoulder. To measure reach, the ulnar styloid process is used as the anatomical landmark. The participant is asked to flexion their shoulder to 90 degrees for the first reading, then to reach as far as possible without any support for the second reading, and finally to return to the starting position. The difference between the two readings is recorded. Each participant is given three trials, and the average is calculated.

SECONDARY OUTCOMES:
Gross grip strength (Jamar hand dynamometer) | Pre-treatment (Week 0) and after treatment (Week 6)
  Standard grip strength is measured using the Jamar hand dynamometer (Pro Med Products, Atlanta, GA) in the standardized test position recommended by the American Society of Hand Therapists, with the patient seated, the arm positioned at the side of the body, and the elbow flexed at 90 degrees. Participants are instructed to squeeze the dynamometer with maximum effort and then fully relax. This procedure is repeated three times for both the right and left hands, and the average values are calculated in kilograms.
Occupational Performance (Canadian Activity Performance Scale (COPM)) | Pre-treatment (Week 0) and after treatment (Week 6)
  The Canadian Occupational Performance Measure (COPM) is a semi-structured, client-centered scale designed to detect changes over time in self-reported occupational performance. It consists of five steps and three scoring phases: (1) The individual identifies occupations in the areas of self-care, productivity, and leisure, rating their importance on a scale from 1 (not important at all) to 10 (extremely important). (2) Using these ratings, the individual selects the five most important occupations. (3) The individual then rates their performance and satisfaction with performance in these selected occupations on a scale from 1 to 10. Two distinct dimensions-Performance and Satisfaction-are evaluated. Each dimension is scored from 1 to 10, with a maximum score of 10 for each. Higher scores indicate better performance and greater satisfaction.
Patient Satisfaction (Patient Satisfaction Short Evaluation Form) | Pre-treatment (Week 0) and after treatment (Week 6)
  The level of patient satisfaction with the treatment they receive is a critical variable for their adherence to treatment and the continuity of their well-being. The scale developed to measure this can yield scores ranging from 0 to 28. Higher scores indicate a greater level of dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: NURGÜL DÜRÜSTKAN ELBAŞI, Study Chair — Istinye University
Locations (1):
- Hüsnü Ayık Care Center, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guideline.

REFERENCES:
- [Background] Cheng C, Liu T, Zhang B, Wu X, Song Z, Zhao Z, Ren X, Zhao M, Su Y, Wang J. Effects of robot-assisted hand function therapy on brain functional mechanisms: a synchronized study using fNIRS and sEMG. Front Med (Lausanne). 2024 Oct 31;11:1411616. doi: 10.3389/fmed.2024.1411616. eCollection 2024. PMID 39544380
- [Background] Zhou Y, Zhao Y, Xiang Z, Yan Z, Shu L, Xu X, Zhang L, Tian X. A dual-task-embedded virtual reality system for intelligent quantitative assessment of cognitive processing speed. Front Hum Neurosci. 2023 Mar 30;17:1158650. doi: 10.3389/fnhum.2023.1158650. eCollection 2023. PMID 37063104
- [Background] Chiaravalloti ND, Weber E, Wylie G, Dyson-Hudson T, Wecht JM. The impact of level of injury on patterns of cognitive dysfunction in individuals with spinal cord injury. J Spinal Cord Med. 2020 Sep;43(5):633-641. doi: 10.1080/10790268.2019.1696076. Epub 2019 Dec 20. PMID 31859606